CLINICAL TRIAL: NCT04814576
Title: Impact of a Collaborative Nursing Care-based Intervention on the Recovery Process, the Therapeutic Relationship, and Positive Mental Health of Day Hospital Users: a Mixed Methods Study Protocol
Brief Title: Collaborative Nursing Care-based Intervention in Mental Health Day Hospital Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FIDMAG Germanes Hospitalàries (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Principal Investigator, Ana Ventosa Ruiz, Mental health nurse, FIDMAG Germanes Hospitalàries
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: CNCMM
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Care Acceptor, Health; Nurse's Role; Relationship, Nurse Patient; Mental Health Disorder; Mental Health Wellness 1
Keywords: Collaborative care; nursing; recovery; therapeutic relationship; positive mental health; participatory action research
MeSH Terms: conditions — Patient Acceptance of Health Care; Mental Disorders

STUDY DESIGN:
Intervention Model Description: A sequential and transformative mixed methods design is proposed.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Collaborative nursing care
  Interventions: Behavioral: Collaborative cares
- Group 2 (No Intervention): Traditional nusing care

INTERVENTIONS:
Behavioral: Collaborative cares — The intervention consists of the co-design and implementation of therapeutic activities by the nurse and the mental health day hospital users following a collaborative care model. For this purpose, the participatory action research (PAR) method will be used and semi-structured interviews and focus groups will be used as data collection techniques.
  Other Names: Co-designing and implementing activities through collaborative nursing care in mental health day hospitals.
  Arms: Group 1

SUMMARY:
OBJECTIVES: 1. To evaluate the impact of an intervention based on collaborative nursing care in terms of the changes produced in the recovery process, in positive mental health and in the nurse-patient therapeutic relationship among users of mental health day hospitals. To explore the changes produced in the recovery process of users who receive collaborative nursing care through the co-design and implementation of group activities.

DESIGN: A sequential and transformative mixed methods design is proposed.

METHODS. The study is structured in three phases. In phase one (baseline) and phase three (follow-up), quantitative data will be collected from patients at a mental health day hospitals based on a two-armed, parallel-design, non-randomized trial. In phase two, two groups will be established: an intervention group (GI) in which the intervention based on collaborative nursing care will be carried out through the co-design and implementation of activities through Participatory Action Research, and a control group (CG) in which the usual care dynamics will be continued. All the users of three mental health day hospitals who agree to participate in the study will be studied consecutively until the necessary sample size is reached. The outcomes used to evaluate the impact of the intervention will be the stage of the recovery process, the quality of the therapeutic relationship and the patient's level of positive mental health.

DISCUSSION: Very few collaborative nursing care interventions have been studied and shown to be effective in the context of the paradigm shift toward recovery in mental health nursing.

IMPACT: Understanding the changes produced in the recovery process, as well as in the quality of the therapeutic relationship and in the maintenance and/or increase of the levels of positive mental health of people with mental health problems, can contribute to the design and implementation of new methodologies to offer effective and person- centered care.

DETAILED DESCRIPTION:
1. Aims A.evaluate the impact of a collaborative nursing care intervention through the co-design and implementation of group activities, in mental health day hospital users, in terms of the changes produced in the state of the recovery process, in the level of positive mental health and in the level of therapeutic relationship with the nurse.

   B. explore the changes produced in the recovery process of mental health day hospital users who receive collaborative nursing care through the co-design and implementation of group activities.

   The research hypotheses to be tested in this study are:

   A. day hospital users who receive an intervention based on collaborative nursing care through the co-design and implementation of group activities will report improved changes in: i) recovery status, ii) level of Positive Mental Health and iii) quality of the therapeutic relationship at the end of the intervention, than users receiving usual care.

   B. the effects of the intervention based on collaborative nursing care through the co-design and implementation of group activities on the changes in the level of recovery are mediated by the changes produced in the quality of the therapeutic relationship and the changes in the positive mental health of the users.
2. Design In order to meet the main objectives, a sequential and transformative mixed methods design is proposed through three phases. On the one hand, in phases 1 and 3, a two-armed, parallel-design, non-randomized trial is proposed. And in phase 2, the intervention will be carried out based on collaborative nursing care through the co-design and implementation of group activities using the qualitative Participatory Action Research (PAR) method.

   2.1. The Participatory-Action Research In order to carry out the intervention of co-design and implementation of activities through collaborative nursing care, PAR is a method that provides a suitable framework for implementation and evaluation, since it is a method that makes it possible to extract knowledge in a democratic, cooperative, transparent and effective way, as well as to intervene in changes in people's daily lives. It is about unveiling the complexity of problems through dialogue and collaboration, as well as acting as a tool to promote change . The PAR process is considered open, holistic and egalitarian, i.e. it equates the researcher with those being researched and requires collaboration between researcher and researched . In general, the PAR consists of four stages that follow each other in a cyclical manner. The cycle begins in the first stage, where a situation or problem is analyzed, and then in the second stage the elements that facilitate its resolution and those that hinder it are identified. Once these factors have been identified, a plan of action or change is developed and implemented. Finally, the effect of this change will be evaluated, thus completing the cycle. All these stages should be evaluated in a reflective manner to improve the rationality, justification and understanding of the changes that occur in the process. In other words, in this PAR process, theory and practice are combined, bringing theoretical constructs into reality and analyzing them simultaneously. Among the different PAR modalities, we will use the one described by Susman and Evered where a process of constant cycles of action research takes place, since it is the one that best adapts to the actual practice of care in the mental health day hospital.
3. Study setting and participants The scope of the study will be three adult mental health day hospitals in the metropolitan area of Barcelona (Spain). The three centers belong to the same institution and are part of the public mental health network of Catalonia. These centers have the same management, and therefore develop the same care program. The study population will be the users requiring treatment in the mental health day hospitals included in the study.

Criteria for selection and recruitment of participants:

- The criteria for inclusion in the study of participating users will be: A) Users over 18 years of age of the selected day hospitals. B) Acceptance of the study conditions and informed consent.

- The exclusion criteria for participating users will be: A) Hospital admission for a period of less than one week. B) Physical or psychological conditions that do not allow collaborative nursing care through co-design of group activities.

All persons who meet the inclusion and exclusion criteria and who agree to participate in the study will be invited. Participants will be incorporated consecutively as they are hospitalized in the three units that form part of the study. To calculate the sample size necessary to have sufficient statistical power for the quantitative part and based on the results of Lemos-Giráldez, accepting an alpha risk of 0.05 and a beta risk of 0.2 in a bilateral contrast, 76 participants would be required in the first group receiving the intervention and 76 in the second group, in order to detect a difference equal to or greater than 5 units. It is assumed that the common standard deviation is 11 and the correlation coefficient between the initial and final measurement is 0.6. A 20% loss-to-follow-up rate was estimated.

4 Procedure, techniques and analysis for the qualitative part or intervention: 4.1 The intervention Given the clinical practice conditions of the study, the intervention will be carried out in the selected hospital using the Participatory Action Research method and will be implemented through a cycle of four well-defined stages which will be repeated continuously throughout the process . Thus, for each user who joins the study, a minimum of one complete cycle will be performed before the user is discharged. The start of the cycle will begin with stage 1 or diagnosis, which will be performed at the time of admission to the day hospital. The nurse, through an individual semi-structured interview, will explore the meaning for the user of the concept of recovery together with the individual perception of the facilitating and limiting elements of this process. Subsequently, in the second stage or planning stage, through a discussion group with other users, the meaning of recovery, as well as its limitations and facilitators will be discussed collectively, whereby individual or collective action plans will be shared by the users in order to work and improve their level of recovery in stage 3 or the action stage. Once the action plan agreed upon by the users and the nurse has been carried out, the cycle will conclude with stage 4 or evaluation, where an individual intervention in the form of a semi-structured interview will be carried out again to assess the recovery process.

4.2 Qualitative data collection techniques Semi-structured interview The conversation will be recorded with the prior consent of the participant and then a written transcript will be prepared, which requires validation by the user to avoid possible biases. The interview should take place in a room, if possible without interruptions and with an approximate duration of 40 minutes. The user will be given the possibility of ending the interview at any time as desired. A script will be used to conduct the interview.

Focus groups These will also be recorded, thanks to the prior consent given by the users. A weekly group will be held at the day hospital's facilities, during the day hospital's hours of operation. It will last approximately 45 minutes. There will be the possibility of leaving the group if the user wishes to do so. To carry out the group, a support script will be followed.

Researcher's diary As a reflective tool and in order to monitor the research process, a field diary written by the principal investigator will be kept.

4.3 Qualitative data analysis The qualitative content analysis method will be used. The data obtained from both the focus groups and the interviews will be transcribed verbatim. Then, once the authenticity of the transcripts has been verified by the participants (content validation), the text will be broken down into descriptive codes assigned on the basis of their purely semantic content. In a second stage, such codes will be grouped into more analytical subcategories, in such a way that the initial codes are grouped according to the meaning of the linguistic units and their combinations. This will lead to a third hierarchical stage, where, taking into account the semantic analysis of the previous subcategories, they will be categorized according to the objectives of the study. It is worth mentioning that the data analysis will be performed by two researchers, jointly in the first stage of data coding, and independently during the subsequent analytical process and again together in the comparison of their results. The analysis of these data will be carried out through the QRS Nvivo v12 program. It should be noted that data will be collected and analyzed qualitatively until the moment when the team considers that no new meanings are found and considers that data saturation has been reached.

3.4 Outcome measures, data collection procedure and data analysis for quantitative phases 4.1 Outcomes Primary outcome Changes in the users' recovery process will be evaluated with The Stages of Recovery Instrument (STORI), validated in the Spanish population by Lemos-Giráldez. It is a self-report questionnaire of 50 items grouped into 5 dimensions of 10 items. Each dimension is related to one of the recovery processes (moratorium, awareness, preparation, rebuilding and growth). The items are scored from 0 "not true at all at this time" to 5 "completely true at this time", resulting in a score for each stage, ranging from 0 to 50. The participant is assigned to the stage with the highest score. The questionnaire has been validated in the Spanish population, obtaining a Cronbach's alpha of 0.86 .

Secondary outcomes The quality of the therapeutic relationship between nurses and users will be evaluated with the Working Alliance Inventory-Short (WAI-S) scale. The short version of this scale contains 12 items, and each item is assessed by the health professional based on a scale ranging from 1 (never) to 7 (always). The scoring range of the overall WAI-S is 12-84 points. The higher the score, the higher the therapeutic relationship. This questionnaire has three dimensions: (i) bond: the bond between patient and nurse, which includes aspects such as empathy, mutual trust and acceptance; (ii) objectives: the agreement between patient and nurse on the goals of therapy (i.e. mutual acceptance of what the intervention aims to achieve); and (iii) tasks or activities: the agreement between patient and nurse on the tasks or activities to be carried out. The Spanish version of the WAI-S has good reliability and validity, with a Cronbach alpha of 0.93 .

The level of positive mental health will be assessed with the Salud Mental Positiva (SMP) scale (Positive Mental Health), developed and validated by Lluch which studies the level of positive mental health, a concept previously developed by Jahoda. The scale consists of 39 scorable items, for which the lowest value is "always or almost always" and the highest value is "never or almost never". The items belong to six dimensions (personal satisfaction, prosocial attitude, self-control, autonomy, problem solving and self-actualization, and interpersonal relationship skills). The questionnaire has shown adequate internal consistency values in different populations with Cronbach's alpha values of 0.89 .

Other outcomes Sociodemographic variables were gathered, including age, sex, educational level, employment status and marital status.

The clinical variables consisted of the main diagnosis described by ICD10 criteria, years of evolution of the disorder, referral unit, number of previous admissions to mental health facilities.

4.2 Data collection procedure Users who agree to participate in the study and have signed the informed consent form, both in the case of the intervention and control groups, will be given a form containing a questionnaire with sociodemographic and clinical data and the three evaluation instruments by a member of the research team who is not directly involved in the care of the users. Participants will not receive any information about their inclusion in the intervention or control group. Each user will be assigned a participant code to ensure the anonymity of the participating users. When the user is discharged, a person from the research team will collect the follow-up data in the same way by means of a new form.

4.3 Quantitative data analysis The principal investigator will construct a database using the IBM SPSS v25 program ECPHDSM, the data obtained from the forms will be incorporated into the database by two members of the research team to minimize error. The analysis will focus on the numerical differences obtained through the STORI, WAI-S and SMP questionnaires before and after the intervention. In order to describe the characteristics of the participants and the scores obtained on the scales, descriptive statistics will be used, using the arithmetic mean and standard deviation for quantitative variables, and the frequency and percentage for qualitative variables. The differences between the baseline scores obtained and the follow-up assessment will be estimated thanks to the application of parametric tests (Student's t-test in paired data) in the case of quantitative variables, first verifying the assumptions of normality and homogeneity of their variances. When the opposite is true, nonparametric tests will be used, using the Wilcoxon test for quantitative variables and Chi-square tests or Fisher's exact test for qualitative variables. In addition, to analyze the impact of changes on the dependent variable adjusted for the remainder of the secondary outcomes, multiple linear regression models will be used. A significance level of p<0.05 will be considered.

5 Ethical considerations Authorization has been obtained from the management of the centers and approval for the project has been granted by the Ethics Committee of the institution where the study will be carried out. In relation to the current law on personal data protection and guarantee of digital rights, the authorization of all users will be requested for the public dissemination of the data, preserving the confidentiality and anonymity of their identity at all times. This will be achieved by anonymizing the names or any sign of identity by assigning a user code. All participants will be able to voluntarily withdraw from the study at any time. For this reason, users will be given a sheet with all the precise information about the study to be carried out and written consent will be requested.

6 Validity and reliability / Rigor To ensure the validity and rigor of the study, appropriate strategies will be used for each phase of the research. In phases 1 and 3, the selection of participants and recruitment of an appropriate sample size together with the validity and reliability of the instruments used will guarantee validity and reliability. For phase 2, reliability, authenticity and ethical criteria will be addressed. Within the framework of reliability, the credibility of the study is based on the use of triangulation of techniques and researchers. Likewise, the criterion of dependence will be obtained through the constant auditing and transfer of external reports throughout the procedure. Likewise, the dynamics of the process, which will involve a constant interaction between the realities of researchers and participants, will provide authenticity to the data obtained. The treatment of confidentiality, privacy and participant consent will guarantee the ethical rigor criteria of the project. In addition, reflexivity, understood as a process of critically reflecting on what is taking place during the research study, will be the key quality criterion upon which the project will be based.

ELIGIBILITY:
Inclusion Criteria:

Users over 18 years of age of the selected day hospitals. Acceptance of the study conditions and informed consent.

Exclusion Criteria:

Hospital admission for a period of less than one week. Physical or psychological conditions that do not allow collaborative nursing care through co-design of group activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Recovery | Two months
  Changes in the users' recovery process will be evaluated with The Stages of Recovery Instrument (STORI) It is a self-report questionnaire of 50 items grouped into 5 dimensions of 10 items. Each dimension is related to one of the recovery processes (moratorium, awareness, preparation, rebuilding and growth). The items are scored from 0 "not true at all at this time" to 5 "completely true at this time", resulting in a score for each stage, ranging from 0 to 50. The higher the score, the better the state of recovery.

SECONDARY OUTCOMES:
Therapeutic relationship | Two months
  The quality of the therapeutic relationship between nurses and users will be evaluated with the Working Alliance Inventory-Short (WAI-S) scale.
  The short version of this scale contains 12 items, and each item is assessed by the health professional based on a scale ranging from 1 (never) to 7 (always). The scoring range of the overall WAI-S is 12-84 points. The higher the score, the higher the therapeutic relationship.
Positive mental health | Two months
  The level of positive mental health will be assessed with the Salud Mental Positiva (SMP) scale (Positive Mental Health) The scale consists of 39 scorable items, for which the lowest value is "always or almost always" and the highest value is "never or almost never". Scores range from 39 to 156. The higher the score, the higher the positive mental health

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Moreno Poyato, Study Director — Universitat de Barceona
Locations (1):
- Benito Menni CASM, Sant Boi de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teddlie, C., & Tashakkori, A. (2012). Common "Core" Characteristics of Mixed Methods Research: A Review of Critical Issues and Call for Greater Convergence. American Behavioral Scientist, 56(6), 774-788.
- [Background] Baum F, MacDougall C, Smith D. Participatory action research. J Epidemiol Community Health. 2006 Oct;60(10):854-7. doi: 10.1136/jech.2004.028662. PMID 16973531
- [Background] Abad Corpa, E., Delgado Hito, M., & Cabrero García, J. (2010). La investigación-acción-participativa: una forma de investigar en la práctica enfermera. Investigación y Educación En Enfermería, 28(3), 464-474.
- [Background] Lavoie, L., Laurin, P., & Marquis, D. (1996). La recherche-action : théorie et pratique : manuel d'autoformation. Presses de l'Université du Québec.
- [Background] Susman, G. I., & Evered, R. D. (1978). An Assessment of the Scientific Merits of Action Research. Administrative Science Quarterly, 23(4), 582. https://doi.org/10.2307/2392581
- [Background] Lemos-Giraldez S, Garcia-Alvarez L, Paino M, Fonseca-Pedrero E, Vallina-Fernandez O, Vallejo-Seco G, Fernandez-Iglesias P, Ordonez-Camblor N, Solares-Vazquez J, Mas-Exposito L, Barajas A, Andresen R. Measuring stages of recovery from psychosis. Compr Psychiatry. 2015 Jan;56:51-8. doi: 10.1016/j.comppsych.2014.09.021. Epub 2014 Oct 18. PMID 25444077
- [Background] Crowe M, Inder M, Porter R. Conducting qualitative research in mental health: Thematic and content analyses. Aust N Z J Psychiatry. 2015 Jul;49(7):616-23. doi: 10.1177/0004867415582053. Epub 2015 Apr 21. PMID 25900973
- [Background] Jayasekara RS. Focus groups in nursing research: methodological perspectives. Nurs Outlook. 2012 Nov-Dec;60(6):411-6. doi: 10.1016/j.outlook.2012.02.001. Epub 2012 Mar 29. PMID 22464693
- [Background] Andrade-González, N., & Fernández-Liria, A. (2016). Spanish Adaptation of the Working Alliance Inventory-Short (WAI-S). Current Psychology, 35(1), 169-177. https://doi.org/10.1007/s12144-015-9365-3
- [Background] Lluch Canut, M. T. (1999). Construccion De Una Escala Para Evaluar La Salud Mental Positiva. In Construccion De Una Escala Para Evaluar La Salud Mental Positiva. Universitat de Barcelona.
- [Background] Jahoda, M. (1959). Current Concepts of Positive Mental Health. The American Journal of Nursing, 59(2), 263. https://doi.org/10.2307/3417722
- [Background] Roldan-Merino J, Lluch-Canut MT, Casas I, Sanroma-Ortiz M, Ferre-Grau C, Sequeira C, Falco-Pegueroles A, Soares D, Puig-Llobet M. Reliability and validity of the Positive Mental Health Questionnaire in a sample of Spanish university students. J Psychiatr Ment Health Nurs. 2017 Mar;24(2-3):123-133. doi: 10.1111/jpm.12358. Epub 2017 Feb 1. PMID 28150373
- [Derived] Ventosa-Ruiz A, Moreno-Poyato AR, Canete-Masse C, Roldua-Ros J, Feria-Raposo I, Campoverde K, Puig Llobet M. Impact of Collaborative Nursing Care on Health Outcomes of Mental Health Day Hospital Users: A Mixed Methods Study. J Psychiatr Ment Health Nurs. 2025 Jun;32(3):575-590. doi: 10.1111/jpm.13133. Epub 2024 Nov 11. PMID 39526836
- [Derived] Ventosa-Ruiz A, Moreno-Poyato A, Lluch-Canut T, Vaquerizo-Cubero A, Vidal-Pascual X, Gil-Guinon F, Puig-Llobet M. Impact of collaborative nursing care on the recovery process of mental health day hospital users: a mixed-methods study protocol. BMJ Open. 2022 Mar 30;12(3):e057969. doi: 10.1136/bmjopen-2021-057969. PMID 35354640